CLINICAL TRIAL: NCT06066411
Title: The Effect of Massage Ball Application on Arterial Blood Pressure, Fatigue and Anxiety in Pregnant Women Diagnosed With Preeclampsia
Brief Title: The Effect of Massage Ball Application on Blood Pressure, Fatigue and Anxiety in Pregnant With Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Filiz Ünal Toprak, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SBU-EBE-ZB-01
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Midwifery; Arterial Blood Pressure; Anxiety; Fatigue
MeSH Terms: conditions — Pre-Eclampsia; Anxiety Disorders; Fatigue

STUDY DESIGN:
Intervention Model Description: Two groups with a massage ball group and control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the application will be performed by the researcher, patients will be blinded in this study. The statistician will be blinded in the evaluation of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage Ball Group (Experimental): A massage ball will be applied to the patients' hands and feet for 20 minutes.
  Interventions: Other: Massage Ball
- Control Group (No Intervention): No application will be made to this group by the researcher.

INTERVENTIONS:
Other: Massage Ball — The massage ball application will be applied to the patients by the researcher for 20 minutes every day for 3 days.
  Arms: Massage Ball Group

SUMMARY:
The aim of this study is to determine the effect of massage ball application on arterial blood pressure, fatigue and anxiety in pregnant women diagnosed with preeclampsia.

DETAILED DESCRIPTION:
Hypertensive disorders are one of the common disorders in pregnancy that cause complications in the mother and the fetus. Preeclampsia, one of the hypertensive disorders of pregnancy, is defined as the presence of hypertension, proteinuria or organ damage that occurs after the 20th week of pregnancy. Preeclampsia affects 5% to 7% of all pregnancies. It causes more than 70,000 maternal deaths and 500,000 fetal deaths worldwide each year. Preeclampsia is among the main causes of maternal mortality and morbidity. Preeclampsia is the first cause of maternal death due to hypertension. According to the report on causes of maternal death in our country, 14.2% of pregnant women died due to hypertensive diseases in 2019. Pregnancy-induced hypertension is the second leading cause of maternal deaths. Preeclampsia causes increased blood pressure in pregnant women, cardiovascular diseases, cerebrovascular accidents, and dysfunction in organs such as the liver, kidney and uterus. In addition to affecting the systems, it is also a condition that causes anxiety and fatigue in pregnant women. The most effective treatment for preeclampsia is delivery. In hospital, treatment includes MgSO4 therapy, blood pressure monitoring, urine monitoring, a high-protein and salt-restricted diet, and control of fetal movements and midwifery care to keep blood pressure at normal levels and prevent eclampsia. In addition to medical treatment in preeclampsia, complementary treatments such as music therapy, acupuncture and massage are also used. Massage application helps relax the muscles. It is stated that massage applied to pregnant women positively affects anxiety, blood pressure and fatigue. Equipment such as tennis ball, golf ball and massage ball are used for muscle relaxation. It is thought that massage ball application, one of the methods used in massage, will reduce anxiety, fatigue and be effective in lowering blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* In the 20th - 40th week of pregnancy,
* Least literate,
* Does not have any diagnosed problems related to fetal health,
* Diagnosed with preeclampsia,
* Will be hospitalized for at least 3 days,
* Not having any physical or mental disability,
* Those who are over 18 years of age,
* Agreeing to participate in the research,
* Women with loss of sensation/sensation,

Exclusion Criteria:

* Those with chronic hypertension,
* Diagnosed with eclampsia,
* Those with HELLP findings,
* Hospital stay of less than 3 days,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since it is a study conducted on pregnant women, it concerns the female gender.
Enrollment: 66 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Arterial Blood Pressure Monitoring Form I-II | Three Days
  They are two separate forms created to evaluate the arterial blood pressure of the pregnant women in the experimental and control groups. Form I was created to evaluate the arterial blood pressure of the pregnant women in the experimental group, and Form II was created to evaluate the arterial blood pressure of the pregnant women in the control group. Form I was created to evaluate the arterial blood pressure of the pregnant women in the control group. In Form I, just before the massage ball application, massage The arterial blood pressure of the pregnant woman was measured for 3 days, 30 minutes, 60 minutes and 90 minutes after the application of the ball. In Form II, unlike Form I, arterial blood pressure measurements are made at the first encounter with the pregnant woman, 30 minutes, 60 minutes and 90 minutes later, without any intervention.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory(STAI) | Three Days
  Each item in the State Anxiety Inventory consists of a four-point Likert scale: Not at all (1), Somewhat (2), Fairly (3), Completely (4), which determines the intensity of the emotions felt by individuals at that moment.
  Each item consists of four options, depending on the frequency of emotions: Almost never (1), Sometimes (2), Often (3), Almost always (4). There are 20 items in each subscale, and 40 items in total. When calculating the State Anxiety Inventory, scoring is done in reverse for items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. The total score obtained from both scales in the inventory varies between 20-80. High scores from the scales indicate high anxiety, while low scores indicate low anxiety levels.
Visual Similarity Scale for Fatigue | Three Days
  It has 2 sub-dimensions: Fatigue and Energy. The 1st, 2nd, 3rd, 4th, 5th, 11th, 12th, 13th, 14th, 15th, 16th, 17th, 18th items of the scale are fatigue and the 6th, 7th, 8th items are fatigue. , 9th and 10th items belong to the energy sub-dimension. It consists of lines with the most positive expression at one end and the most negative expression at the other end, with 10 cm lines between the two expressions.
  Individuals are asked to mark the part that is suitable for them on a 10 cm line. Then, the value is determined by measuring the marked part with a ruler. While the fatigue subscale items go from the most positive to the most negative, the energy subscale items go from the most negative to the most positive. A high score from the fatigue sub-dimension and a low score from the energy sub-dimension indicates that the severity of fatigue is high.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Bicav, Principal Investigator — Saglik Bilimleri Universitesi; Filiz Ünal Toprak, PhD, Principal Investigator — Saglik Bilimleri Universitesi; Şevki Çelen, PhD, Principal Investigator — Ankara Etlik Şehir Hastanesi
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No